CLINICAL TRIAL: NCT01817608
Title: Weaning From Mechanical Ventilation in the ICU
Status: Completed | Type: Observational
Sponsor: Amal Jubran (Other)
Responsible Party: Sponsor-Investigator, Amal Jubran, Faculty, Loyola University
Organization: Loyola University (Other)
Other Study IDs: 107589
Record Dates: First submitted 2013-03-15; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Quality of Life
Keywords: sf-36; Katz

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators objective is to assess quality of life and functional outcome in patients requiring short-term mechanical ventilation. Additionally, the investigators plan to measure the recovery of peripheral muscle strength and respiratory muscle strength during recovery.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who require mechanical ventilation for at least 2 days
* the ability to speak English
* willing to participate

Exclusion Criteria:

* patients who require mechanical ventilation at home before hospitalization
* patients previously requiring mechanical ventilation at an LTAC facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients receiving mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2004-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
quality of life scores | up to one year after discharge
  SF-36, Katz, respiratory muscle strength and handgrip strength will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Amal Jubran, MD, Principal Investigator — Loyola Univ Chicago Health Sciences Division
Locations (1):
- Loyola University Chicago Health Sciences Division, Maywood, Illinois, United States